CLINICAL TRIAL: NCT01638858
Title: A Prospective, Non-randomized, Mono-center, Cohort Study of Evaluate the Effects of 0.5mg Intraocular Ranibizumab (Lucentis)Injections on Retinal Function in Patients With Diabetic Macular Edema (DME) During Twelve Months
Brief Title: Treatment of Diabetic Macular Edema With 0.5mg Intraocular Ranibizumab (Lucentis)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Dr. Matthias Lueke, Principal Investigator, University of Luebeck
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Lucentis_DME_ERG; 2011-002202-70 (EudraCT Number)
Record Dates: First submitted 2012-07-02; First posted 2012-07-12 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Ranibizumab

ARMS (1):
- Lucentis (Ranibizumab) (Experimental)
  Interventions: Drug: Lucentis (Ranibizumab)

INTERVENTIONS:
Drug: Lucentis (Ranibizumab) — Ranibizumab Short- and Log-term Effects on Retinal Function measured by Multifocal-ERG and Microperimetry

SUMMARY:
In this prospective, open-label clinical study is to investigate the behavior of the retinal functions during development of diabetic macular disease (DME) under the influence of Lucentis. Measurements with the multifocal electroretinogram (ERG) and microperimetry is used here as an objective criteria to information about the retinal function obtain.

ELIGIBILITY:
Inclusion Criteria:

1. diabetic macular edema with center involvement in at least one eye
2. patients with a central retinal thickness
3. patients with a BCVA of 78-24 EDTRS letters
4. decrease in vision is due to DME and not due to other causes, in the opinion of the investigator
5. Type 1 or type 2 diabetes mellitus diagnosed 2 years prior to screening

Exclusion Criteria:

1. history or evidence of severe cardiac disease
2. clinical or medical history uncontrolled hypertension or diabetes
3. of unstable angina, acute coronary syndrome, myocardial infarction or revascularization with 6 months
4. ventricular tachyarrhythmias requiring ongoing treatment
5. history or evidence clinically significant peripheral vascular disease, such a intermittent claudication or prior amputation
6. clinically significant impaired renal or hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-10; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Main outcome measures are the changes of retinal function of the macula monitored by multifocal-ERG as measured 12 months | 12 months
  Main outcome measures are the changes of retinal function of the macula monitored by multifocal-ERG as measured 12 months

SECONDARY OUTCOMES:
to document changes in best corrected visual acuity measured on 4 meters | 12 months
  to document changes in best corrected visual acuity measured on 4 meters
to document changes in microperimetry | 12 months
  to document changes in microperimetry
to document changes in optical coherence tomography (OCT) | 12 months
  to document changes in optical coherence tomography (OCT)

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Grisanti, M.D. Prof., Principal Investigator — University of Luebeck - Department of Ophthalmology: Germany
Locations (1):
- University of Luebeck - Department of Ophthalmology, Lübeck, Germany

REFERENCES:
- See also: Link Text: University of Lübeck - Department of Ophthalmology - Germany — http://www.uksh.de/Augenklinik_Lübeck/index.html